CLINICAL TRIAL: NCT01172834
Title: The Possible Influence of Health Promotion Coaching on Health Related and Organizational Outcomes Among Nurses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Izthak Shapira MD, Tel-Aviv Sourasky Medical Center, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: TASMC-09-IS-0258-09-TLV-CTIL
Record Dates: First submitted 2010-07-18; First posted 2010-07-30 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-07

CONDITIONS: Healthy
Keywords: Nurses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling (Experimental)
  Interventions: Behavioral: Health Coaching

INTERVENTIONS:
Behavioral: Health Coaching — A manual-driven group Health Coaching intervention. Once a week for 3 months.

SUMMARY:
Strong evidence shows that physical activity (PA) has favorable psychological and health related outcomes. However, most employees do not perform enough PA to achieve health and well being benefits. Worksite interventions aimed at improving PA often yield modest effect sizes, and their theoretical ground is not profound. The Health Action Process Approach (HAPA), is a novel comprehensive theoretical model for health behavior change, that hasn't been studied as a whole in a worksite intervention study.

The objectives of the proposed study are:

1. To develop a coaching-based group intervention that will be both grounded in theory (HAPA) as well as applicable.
2. To evaluate the feasibility of conducting this intervention among employed hospital nurses, using a randomized controlled design, interviews and other evaluation procedures.

The proposed study will offer the most comprehensive empirical test to date of the full HAPA model.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working in a full time capacity at Tel-Aviv Sourasky Medical Center.

Exclusion Criteria:

* None nurses or nurses working part-time at Tel-Aviv Sourasky Medical Center.
* Nurses not working at Tel-Aviv Sourasky Medical Center.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-08 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Metabolic Syndrome Ratings | Time 0
  (Blood pressure, Sugar levels, HDL, Triglycerides, Weight)
Metabolic Syndrome Ratings | Time 1 - 3 months Follow up
  (Blood pressure, Sugar levels, HDL, Triglycerides, Weight)
Metabolic Syndrome Ratings | Time 2 - 6 Months Follow up
  (Blood pressure, Sugar levels, HDL, Triglycerides, Weight)
Metabolic Syndrome Ratings | Time 3 - 9 Months Follow up
  (Blood pressure, Sugar levels, HDL, Triglycerides, Weight)

SECONDARY OUTCOMES:
Organizational Behavior Ratings | Time 0
  Absenteeism,Perceived Organizational Support, Organizational Cynicism, Vigor, exhaustion, Peer Support, Social networks
Psychological Ratings | Time 0
  Subjective Well-Being, Psychological Well-Being, Positive and Negative Affect, Self Efficacy, HAPA Stage
Demographic ratings | Time 0
  Age, Gender, Seniority, Marital Status, Number of Kids
Coaching Process Ratings | Time 0
  Goal Attainment
Organizational Behavior Ratings | Time 1 - 3 months follow up
  Absenteeism,Perceived Organizational Support, Organizational Cynicism, Vigor, exhaustion, Peer Support, Social networks
Organizational Behavior Ratings | Time 2 - 6 Months Follow up
  Absenteeism,Perceived Organizational Support, Organizational Cynicism, Vigor, exhaustion, Peer Support, Social networks
Psychological Ratings | Time 1 - 3 months follow up
  Subjective Well-Being, Psychological Well-Being, Positive and Negative Affect, Self Efficacy, HAPA Stage
Psychological Ratings | Time 2 - 6 Months Follow up
  Subjective Well-Being, Psychological Well-Being, Positive and Negative Affect, Self Efficacy, HAPA Stage
Coaching Process Ratings | Time 1 - 3 months follow up
  Goal Attainment
Coaching Process Ratings | Time 2 - 6 Months Follow up
  Goal Attainment
Organizational Behavior Ratings | Time 3 - 9 Months Follow up
  Absenteeism,Perceived Organizational Support, Organizational Cynicism, Vigor, exhaustion, Peer Support, Social networks
Psychological Ratings | Time 3 - 9 Months Follow up
  Subjective Well-Being, Psychological Well-Being, Positive and Negative Affect, Self Efficacy, HAPA Stage
Coaching Process Ratings | Time 3 - 9 Months Follow up
  Goal Attainment

CONTACTS AND LOCATIONS:
Overall Officials: Izthak Shapira, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel